CLINICAL TRIAL: NCT03333252
Title: Dual Target Program: An Non-pharmacological Intervention for Family Caregivers and Patients With Alzheimer's Disease
Brief Title: A Non-pharmacological Intervention for Patients With Alzheimer's Disease and Family Caregivers (Care Partners Program)
Acronym: CPProgram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1803019068; 5R01AG054009 (NIH)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Caregiver
Keywords: Caregiver; Psycho-social intervention; Cognitive training; Quality of life; Early on-set Alzheimer's Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): Exposing caregivers to caregiving-related information and care recipients to cognitive training tasks
  Interventions: Behavioral: Intervention Condition
- Control Condition (Placebo Comparator): Exposing caregivers to Nutrition and Health promotional material. The care recipients are exposed to plain words games from computer.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Intervention Condition — Caregivers will access caregiving related information. Care Recipients will access cognitive training program
  Arms: Intervention Condition
Behavioral: Control Condition — Caregivers will access Nutrition and Health Promotion material. Care Recipients will access words and card games
  Arms: Control Condition

SUMMARY:
The proposed study will develop and test the efficacy and feasibility of a dyadic-based intervention program (DT), delivered through state-of-the art computer tablet technology. A novel feature of the investigation is its focus on both the caregiver and the recipient of care (person with AD) and the integration of an evidenced-based caregiver intervention and evidenced-based cognitive/functional training for the care recipient. The program will be tailored for the caregiver and emphasize issues important to caregivers, not only in the earlier stages of caregiving, but will also target issues across the caregiving trajectory to help prepare the caregiver for changes in their role. Two hundred and forty Hispanic, African American and White/Caucasian dyads will be randomized to the DT intervention or Control condition. Measures at baseline and the 6 and 12-month follow-ups will include indices of care recipient processing speed and quality of life, and caregiver outcomes such as; depression, burden, self-care activities and social support . Information will also be gathered on ethnic differences in response to the intervention and estimates of cost effectiveness of the intervention.

DETAILED DESCRIPTION:
We will recruit and randomly assign, following a baseline assessment, 246 dyads will be enrolled and randomly assigned to one of two groups: 1) Caregiving Condition or 2) Health Promotion (Nutrition) Condition. The entire study is home-based. The intervention will be delivered over 6 months using computer tablet technology in Spanish or English. Assessments will occur in the beginning of the study, 6 months, and 12 months (after completion of the intervention)

Interested participants (caregivers) can contact us via telephone or email after seeing a flyer posted in various WCM/NYP locations including the Irving Sherwood Wright Center on Aging. One of our research associates (RA) will provide more information about the study to potential participants. The trained RA will use a telephone script with consent language to obtain permission to ask them questions to determine their eligibility through a phone screen script. If the participant is ineligible for the study, all screening data will be deleted. If the caregiver participant is eligible for the study, an appointment will be provided, and one of our RAs will visit the participants (caregiver and care recipient) and conduct the baseline assessment at the participants' home in their preferred language (Spanish or English). This assessment with the caregiver will last between 2 and 3 hours, additionally the assessment with the care recipient will last approximately 1.5 hours. We will use Qualtrics (online survey/data collection service) to administer the assessments.

The baseline assessment with the caregiver (CG) consists of a series of questionnaires assessing the level of burden, and depression perceived by the CG while providing the care, the amount of social support available to the CG, and the self-care activities of the CG to provide continuing care to their loved ones. The assessment with the care recipient consists of measures of processing speed (digit symbol). In addition, the care recipient will complete a computer-based questionnaire assessing their quality of life. The assessment with the caregiver and care recipient might not be completed in the same home visit. The study protocol allows multiple visits to complete the assessments.

During the baseline home visit, the RA will go over the written informed consent and HIPAA authorization with the participants (caregiver and care recipient). The assessment will not begin unless the participant has a full understanding of the informed consent form and has signed the form. The care recipient will additionally be given a Consent Feedback Tool, as an added step to make sure they understand the consent form since they have mild cognitive impairment.

ELIGIBILITY:
CAREGIVER (CG)

Inclusion Criteria:

* MMSE ≥ 26 (with Mungus age and education correction)
* Providing care for a friend or relative with AD for a minimum of eight hours per week for at least the past six months
* Being over the age of 21 years
* Living with or nearby the patient
* Having a telephone
* Planning to stay in the study geographic area for the duration of the study

Exclusion Criteria:

* Not providing care to someone with memory problems
* Paid caregivers
* Has terminal illness with life expectancy of 6 months or less

CARE RECIPIENT (CR)

Inclusion Criteria:

* MMSE 18 - 25 (with Mungus age and education correction) (if scores high on MMSE, the care recipient has to score 1.0 in the Clinical Dementia Rating Scale (CDR))
* Needs help with higher level of IADL (e.g., managing finances, helping remember appointments, handling medications)
* Show memory problems

Exclusion Criteria:

* Lives in nursing home or facility
* Going to be placed in a facility in the next 6 months
* Has terminal illness with life expectancy of 6 months or less

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J. Czaja, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Care Recipients - Intervention Condition: Exposing care recipients to cognitive training tasks.
- Care Recipients - Control: Exposing care recipients to plain words games from computer.
- Caregivers - Intervention Condition: Exposing caregivers to caregiving-related information.
- Caregivers - Control: Exposing caregivers to Nutrition and Health promotional material.
Period: Overall Study
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control | Caregivers - Intervention Condition | Caregivers - Control
Started | 89 | 87 | 89 | 87
Completed | 56 | 45 | 64 | 58
Not Completed | 33 | 42 | 25 | 29
Not completed — Adverse Event | 10 | 6 | 5 | 2
Not completed — Death | 1 | 3 | 0 | 0
Not completed — Lack of Efficacy | 8 | 4 | 0 | 7
Not completed — Lost to Follow-up | 0 | 5 | 9 | 3
Not completed — Withdrawal by Subject | 14 | 24 | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Care Recipients - Control Condition: Exposing care recipients to plain words games from computer.
- Caregivers - Control Condition: Exposing caregivers to Nutrition and Health promotional material.
- Total: Total of all reporting groups
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control Condition | Caregivers - Intervention Condition | Caregivers - Control Condition | Total
Number analyzed (Participants) | 89 | 87 | 89 | 87 | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 43 | 36 | 83
  >=65 years | 88 | 84 | 46 | 51 | 269
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 81 [75 to 86] | 81 [76 to 87] | 65 [58 to 74] | 67 [58 to 75] | 75 [65.25 to 83]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 40 | 34 | 74 | 76 | 224
  Male | 49 | 52 | 15 | 11 | 127
  Other | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 19 | 18 | 72
  Not Hispanic or Latino | 73 | 68 | 70 | 69 | 280
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 5 | 0 | 4 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 7 | 8 | 6 | 7 | 28
  White | 75 | 70 | 77 | 73 | 295
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 2 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 89 | 87 | 89 | 87 | 352
Change in depression score for caregiver as measured by CES-D [Median (Inter-Quartile Range); unit: units on a scale] — CES-D is Center for Epidemiological Studies Depression scale, (range 0-30) higher score indicates greater depression Population: The primary outcome listed in the submission is caregiver specific.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 89 | 87 | 176
    (all) |  |  | 9 [7 to 14] | 10 [7 to 13] | 10 [7 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Score for Caregiver as Measured by CES-D
Description: Higher score on the Center for Epidemiological Studies Depression scale (CES-D) means greater frequency of depressive symptoms. Range (0-30)
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: This measure was only administered to caregivers. Missing data is due to participants either lost to follow up or withdrew between the baseline assessment and 12 month assessment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control Condition | Caregivers - Intervention Condition | Caregivers - Control Condition
Number analyzed (Participants) | 0 | 0 | 89 | 87
units on a scale
  baseline |  |  | 9 [7 to 14] | 10 [7 to 13]
  6 month: number analyzed (Participants) | 0 | 0 | 66 | 64
  6 month |  |  | 9 [6.7 to 12] | 8 [5.5 to 11]
  12 month: number analyzed (Participants) | 0 | 0 | 62 | 57
  12 month |  |  | 9 [6 to 13] | 9 [7 to 12]

2. Secondary Outcome: Change in Caregiving Burden Score for Caregiver as Measured by Burden Inventory
Description: Higher score means greater level of caregiver burden. Range (0-44)
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: This measure was only administered to caregivers. Additionally, missing data is due to some participants either being lost to follow up or withdrew between the baseline assessment and 12 month assessment.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control | Caregivers - Intervention Condition | Caregivers - Control
Number analyzed (Participants) | 0 | 0 | 89 | 87
score on a scale
  Baseline |  |  | 18 [13 to 26] | 18 [12 to 25]
  6 month: number analyzed (Participants) | 0 | 0 | 65 | 64
  6 month |  |  | 16 [9.8 to 22] | 15 [9.4 to 23.5]
  12 month: number analyzed (Participants) | 0 | 0 | 61 | 57
  12 month |  |  | 15.6 [9 to 25] | 17 [11 to 24]

3. Other Pre Specified Outcome: Change in Caregiver's Self Report of Self-care
Description: Higher score means better in keeping medical obligations to him/herself. Range (0-12)
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: This measure was only administered to caregivers. Additionally, missing data is due to some participants being either lost to follow up or withdrew between the baseline assessment and 12 month assessment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control | Caregivers - Intervention Condition | Caregivers - Control
Number analyzed (Participants) | 0 | 0 | 89 | 87
units on a scale
  Baseline |  |  | 6 [4.8 to 8.7] | 6 [4 to 8.4]
  6 month: number analyzed (Participants) | 0 | 0 | 65 | 58
  6 month |  |  | 6.6 [4.8 to 8.4] | 6 [4.8 to 7]
  12 month: number analyzed (Participants) | 0 | 0 | 56 | 52
  12 month |  |  | 8 [6.8 to 8.7] | 8 [6.8 to 9]

4. Other Pre Specified Outcome: Change in Caregiver's Social Support
Description: Higher score means more social support for the caregiver. Range (0-40)
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control | Caregivers - Intervention Condition | Caregivers - Control
Number analyzed (Participants) | 0 | 0 | 89 | 87
units on a scale
  Baseline |  |  | 22 [17.1 to 29] | 23 [18.7 to 29]
  6 month: number analyzed (Participants) | 0 | 0 | 63 | 65
  6 month |  |  | 21 [17 to 28.6] | 23 [17 to 28]
  12 month: number analyzed (Participants) | 0 | 0 | 62 | 57
  12 month |  |  | 21.5 [15 to 27.5] | 22 [16.5 to 26]

5. Other Pre Specified Outcome: Change in Care Recipient's Qualify of Life
Description: Higher score means better quality of life as Alzheimer's patient. Range (0-52)
Time Frame: Baseline, 6-mth follow-up, and 12-mth follow-up
Population: This measure was only administered to care recipients. Additionally, missing data is due to some participants being either lost to follow up or withdrew between the baseline assessment and 12 month assessment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control | Caregivers - Intervention Condition | Caregivers - Control
Number analyzed (Participants) | 87 | 87 | 0 | 0
units on a scale
  Baseline | 33 [29 to 36] | 32 [28.6 to 36] |  |
  6 month: number analyzed (Participants) | 55 | 58 | 0 | 0
  6 month | 33 [29 to 36] | 32 [29 to 36] |  |
  12 month: number analyzed (Participants) | 49 | 42 | 0 | 0
  12 month | 33 [29.3 to 37] | 33 [30 to 36] |  |

6. Other Pre Specified Outcome: Change in Care Recipient's Processing Speed Using Digit Symbol Test
Description: Higher score means faster processing speed. Range (0-100)
Time Frame: Baseline, 6-mth follow-up, and 12-mth follow-up
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control | Caregivers - Intervention Condition | Caregivers - Control
Number analyzed (Participants) | 54 | 47 | 0 | 0
units on a scale
  Baseline | 15 [9 to 28] | 27 [19 to 34] |  |
  6 months: number analyzed (Participants) | 19 | 19 | 0 | 0
  6 months | 25 [14 to 30] | 28 [15 to 31] |  |
  12 months: number analyzed (Participants) | 12 | 9 | 0 | 0
  12 months | 20 [14 to 32] | 23 [13 to 30] |  |

ADVERSE EVENTS:
Time Frame: Five years
Groups:
- Care Recipients - Control: The care recipients are exposed to plain words games from computer.
Arm/Group | Care Recipients - Intervention Condition | Care Recipients - Control | Caregivers - Intervention Condition | Caregivers - Control
All-Cause Mortality (participants affected / at risk) | 1/89 | 3/87 | 0/89 | 0/87
Serious Adverse Events (participants affected / at risk) | 11/89 | 12/87 | 2/89 | 5/87
Other Adverse Events (participants affected / at risk) | 7/89 | 18/87 | 26/89 | 16/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Care Recipients - Intervention Condition (N=89) | Care Recipients - Control (N=87) | Caregivers - Intervention Condition (N=89) | Caregivers - Control (N=87)
Emergency Room Visit (General disorders) | 6 | 7 | 0 | 3
Hospitalized (General disorders) | 2 | 1 | 0 | 1
Driving Impairment (General disorders) | 0 | 1 | 0 | 0
Access to Dangerous Object (General disorders) | 1 | 0 | 0 | 0
Hip Replacement (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Institutionalized (General disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Medical problem (General disorders) | 0 | 1 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Care Recipients - Intervention Condition (N=89) | Care Recipients - Control (N=87) | Caregivers - Intervention Condition (N=89) | Caregivers - Control (N=87)
Self-reported depression (Psychiatric disorders) | 1 | 8 | 26 | 15
Allergic reaction (General disorders) | 0 | 1 | 0 | 0
Broken back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Health problems (General disorders) | 0 | 2 | 0 | 0
Forehead injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Heart condition (Cardiac disorders) | 0 | 1 | 0 | 0
Heart surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 1 | 0
Macular Degeneration (Eye disorders) | 1 | 0 | 0 | 0
Hernia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Knee surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Leg fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT03333252/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03333252/ICF_000.pdf